CLINICAL TRIAL: NCT05267262
Title: A Phase II, Multi-center, Open-Label Study to Assess Safety, Tolerability, Efficacy and Pharmacokinetics of R3R01 in AS Patients With Uncontrolled Proteinuria on ACE/ARB Inhibition and in Patients With Primary Steroid-Resistant FSGC
Brief Title: Study to Evaluate R3R01 in Patients With Alport Syndrome and Patients With Focal Segmental Glomerulosclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: River 3 Renal Corp. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R3R01-ASFSGS-201
Record Dates: First submitted 2022-02-23; First posted 2022-03-04 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Alport Syndrome; Focal Segmental Glomerulosclerosis
Keywords: FSGS; Kidney Disease; glomeruli
MeSH Terms: conditions — Nephritis, Hereditary; Glomerulosclerosis, Focal Segmental; Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 2 (Alport Syndrome Patients) (Experimental): R3R01 administered orally as 200 mg tablets twice daily for 84 days.
  Interventions: Drug: R3R01
- Cohort 3 (Focal Segmental Glomerulosclerosis Patients) (Experimental): R3R01 administered orally as 200 mg tablets twice daily for the 84 days.
  Interventions: Drug: R3R01

INTERVENTIONS:
Drug: R3R01 — R3R01 administered orally for 12 weeks

SUMMARY:
This is a Phase 2, Multi-center, Open-Label Study to Assess Safety, Tolerability, Efficacy and Pharmacokinetics of R3R01 in Alport Syndrome Patients with Uncontrolled Proteinuria on ACE/ARB Inhibition and in Patients with Primary Steroid-Resistant Focal Segmental Glomerulosclerosis

DETAILED DESCRIPTION:
R3R01 is investigational small molecule designed to decrease fat levels in certain cells in the kidney and therefore may improve kidney function and reduce damage in the kidney. This is a single arm open-label study enrolling patients in three cohorts. Cohort 1 will include 5 adult (≥18 y/o) patients from Cohorts 2 and 3 (including at least one patient from Cohort 2 and at least one patient from Cohort 3). Cohort 2 will include approximately 20 male and female patients from 12 years and older with X-linked Alport Syndrome (AS), and male and female patients with autosomal inherited AS. Cohort 3 will include approximately 30 male and female patients from age 12 to 75 years with a biopsy proven diagnosis who present with primary steroid-resistant focal segmental glomerulosclerosis (FSGS) with proteinuria.

All eligible patients will be enrolled to receive R3R01 over a treatment period of 12 weeks with a primary efficacy outcome as the percentage change in proteinuria from baseline to the end of treatment (Day 84) in each cohort as a whole

ELIGIBILITY:
Inclusion Criteria:

All Patients:

1. Patient is able to communicate well with the investigator, understands and is willing to comply with all requirements of the study, and understands and signs the written informed consent form (ICF).
2. For children to be eligible, one or both parents/legal guardians must sign a parental permission form which provides information contained in the ICF. Children capable of assent must express their willingness to participate by signing an assent form.
3. If patient has received a COVID vaccination, the baseline visit must occur at least one week or more after the second/booster vaccination.
4. Patients who have had active symptoms of COVID within 3 months prior to screening and are now asymptomatic for the last 2 weeks but have tested COVID PCR positive. If a patient is asymptomatic at screening but is COVID positive, then rescreening can occur after a minimum of two weeks.
5. Both female patients, as well as, female partners of male patients who are of child-bearing potential must be willing to not become pregnant for the complete duration of the study (>180 days) (90 days after the last dose of study medication).
6. Males (including sterilized subjects) whose female partners have child-bearing potential, must agree to use male contraception (condoms) during the period from the time of signing the informed consent form (ICF) through 90 days after the last dose of study drug. They must agree to immediately inform the investigator if their partner becomes pregnant during the study.

   Alport Syndrome Patients Inclusion Criteria (in addition):
7. Males and females with X-Linked AS and males and females with autosomal inherited AS.

   1. For countries that are enrolling pediatric patients: patients from age 12 years and older.
   2. For countries that are not enrolling pediatric patients: patients from age 18 years and older.
8. Confirmed diagnosis of AS by genetic testing and /or kidney biopsy. For patients enrolled in the US who meet all inclusion and exclusion criteria but have not had their diagnosis confirmed by genetic testing or kidney biopsy, the Sponsor will provide for patient's genetic testing.
9. UPCR ≥1.0 g/g.
10. eGFR ≥ 30 mL/min/1.73m2 (using CKD-EPI equation for adults and Bedside Schwartz equation for children).
11. ACEi/ARB therapy at maximum tolerated dose stable for at least 4 weeks prior to enrollment and during the study.

    Focal Segmental Glomerulosclerosis Patients Inclusion Criteria (in addition):
12. Male or female patients,

    1. For countries that are enrolling pediatric patients: 12 to 75 years old at the time of signing the informed consent
    2. For countries that are not enrolling pediatric patients: 18 to 75 years old at the time of signing the informed consent
13. Primary FSGS, (without any identifiable cause, and where the FSGS is confirmed by renal biopsy) or FSGS where there is documentation of a genetic mutation in a podocyte protein associated with FSGS.
14. If on steroids, the dose should remain stable for at least 4 weeks prior to enrollment and during the study. Subjects who are steroid-resistant, defined as failure to achieve partial or complete remission, or subjects who experienced adverse events without acceptable clinical benefit after at least 8 weeks of adequate corticosteroid therapy for children and 12 weeks for adults are eligible.
15. UPCR between 1.5g/g and 12.0g/g.
16. eGFR > 30 mL/min/1.73m2 (using CKD-EPI equation for adults and Bedside Schwartz equation for children).
17. If taking concomitant ACEi and/or ARB treatment, it should remain at a stable dose for at least 4 weeks prior to enrollment and during the study.

Exclusion Criteria:

All Patients:

1. Uncontrolled diabetes mellitus as evidenced by an HbA1c ≥ 11%. For Germany: HbA1c ≥ 8.5%.
2. Uncontrolled hypertension

   1. Adults: (SBP ≥ 180mmHg and/or DBP ≥ 100mmHg). For Germany: (SBP ≥ 140mmHg and/or DBP ≥ 100mmHg).
   2. Children: ≥ 95th percentile or ≥ 130/80 mm Hg, whichever is lower
3. Moderate or severe hepatic impairment (Child-Pugh B or C), except if (a) decreased serum albumin is directly related to the renal disease (resulting in a Child Pugh score of 7), and (b) no other Child-Pugh Score parameters are increased and (c) patient has no liver pathology in medical history.
4. Presence of any active (i.e., with symptoms) and/or uncontrolled infection (including COVID).
5. Presence of Human immunodeficiency virus (HIV).
6. BMI > 40. Note - For Germany: BMI > 35 (Obesity Class II).
7. History of malignancy other than treated basal cell or squamous cell skin cancer within the past 5 years.
8. History of alcohol abuse in the last 5 years or currently drinks in excess of 21 and 14 units per week for males and females, respectively.
9. Received an investigational agent within 30 days or 5 half-lives prior to screening (whichever is longer).
10. History of non-compliance such that patient is unlikely to be compliant with study visits, procedures or drug administration.
11. Patient has had an organ transplant, is currently on an organ transplant waiting list or there is a reasonable possibility that the patient will have an organ transplant in the 6 months after screening.
12. Participation in an interventional trial within the previous 3 months prior to screening or concurrent participation in a research trial.
13. Patient is not suitable to participate in the study for any reason (including, but not limited to co-morbidities, history of non-compliance with study visits, procedures, or drug administration) in the opinion of the investigator.
14. Females of childbearing potential (those who are not surgically sterilized or post-menopausal for at least 1 year) are excluded from participation in the study unless they agree to use highly effective contraception.
15. Females that are lactating.
16. History of hypersensitivity to study drug and/or any of its excipients.
17. Patients with hereditary galactose intolerance, total lactase deficiency or glucose-galactose malabsorption.
18. Required concomitant use of bardoxolone, rituximab, cyclo-phosphamide, abatacept, or sparsentan

    Alport Syndrome Patients Exclusion Criteria (in addition):
19. Kidney disease apart from AS, e.g. diabetic nephropathy or lupus nephritis.
20. Use of Bardoxolone or sparsentan treatment in the 30 days prior to screening. SGLT2 inhibitors are allowed if the patient is on a stable dose for at least 3 months prior to enrollment and during the study.

    Focal Segmental Glomerulosclerosis Patients Exclusion Criteria (in addition):
21. Patient has collapsing variant of FSGS on renal biopsy.
22. Patient has FSGS secondary to another condition (e.g. obesity, cardiovascular, infectious, or autoimmune disorder).
23. Use of Rituximab, cyclophosphamide or abatacept treatment in the 120 days prior to screening. If taking other chronic immune-modulatory medications that are small molecules, the dosage must be stable for 4 weeks prior to screening and during the study.
24. If previous Rituximab treatment is greater than 120 days from screening, CD20 cell count should be within normal limits.
25. If previous other antibody treatment on a stable dose is greater than 120 days from screening, the investigator must deem administration of study drug to be safe.
26. Use of sparsentan in the 30 days prior to screening. SGLT2 inhibitors are allowed if the patient is on a stable dose for at least 3 months prior to enrollment and during the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2025-05-21 (Actual); Study Completion 2025-08-19 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (Safety and Tolerability) | 12 weeks
  Safety and tolerability as determined by the incidence of adverse events (AEs)
Assess change in urine creatinine protein ratio | 12 weeks
  Change from baseline in urine creatinine protein ratio for Cohort 1 (Alport Syndrome patient group) and Cohort 2(Focal Segmental Glomerulosclerosis patient group).

SECONDARY OUTCOMES:
Change in quality-of-life assessment from baseline to end of treatment and to the end of the follow-up period by cohort for adults | 24 weeks
  Change in quality of life as measured by the Short Form SF-36 for adults
Change in quality-of-life assessment from baseline to end of treatment and to the end of the follow-up period by cohort for children | 24 weeks
  Change in quality of life as measured by the pediatric quality of life inventory (PedsQL) for children

CONTACTS AND LOCATIONS:
Locations (22):
- United States (14):
  - Investigative Site, Los Angeles, California
  - Investigative site, Boca Raton, Florida
  - Investigative site, Miami, Florida
  - Investigative site, Riverview, Florida
  - Investigative site, Atlanta, Georgia
  - Investigative site, Boston, Massachusetts
  - Investigative site, Ann Arbor, Michigan
  - Investigative site, Minneapolis, Minnesota
  - Investigative Site, Cary, North Carolina
  - Investigative site, Cleveland, Ohio
  - Investigative site, Columbus, Ohio
  - Investigative site, East Providence, Rhode Island
  - Investigative Site, Dallas, Texas
  - Investigative site, Houston, Texas
- Belgium (2):
  - Investigative site, Brussels
  - Investigative site, Liège
- Investigative site, Paris, France
- Investigative site, Göttingen, Germany
- Netherlands (2):
  - Investigative site, Amsterdam
  - Investigative site, Nijmegen
- United Kingdom (2):
  - Investigative site, Leicester
  - Investigative site, Nottingham

IPD SHARING:
Plan to Share IPD: No